CLINICAL TRIAL: NCT06734377
Title: Causal Role of Delta and Theta Oscillations in Hierarchical Cognitive Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Justin Riddle, Principal Investigator, Florida State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 00005546
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Rhythmic Transcranial Magnetic Stimulation (rTMS) Effect on Hierarchical Cognitive Control
Keywords: Rhythmic Transcranial Magnetic Stimulation; Hierarchical Cogntive Control

STUDY DESIGN:
Intervention Model Description: Each participant receives all three types of stimulations (delta, theta, arrhythmic) in both brain regions, with the order of stimulation randomized for each session. Across the 12 task blocks in each session with the stimulation, the type of stimulation is interleaved, ensuring that all conditions are represented in a balanced manner. The number of trials for each stimulation condition is counterbalanced within and across blocks to provide equal exposure to each type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TMS to Mid-dlPFC followed by TMS to PMd (Experimental): Participants would receive TMS while performing a cognitive control task. In their first stimulation session, the TMS coil will be placed over mid-dlPFC region on the scalp. In their second session, the TMS coil will be placed over the PMd region on the scalp. During every session, participants receive Delta TMS (2.2 Hz), Theta TMS (6.5 Hz), and Arrhythmic TMS.
  Interventions: Device: Delta TMS; Device: Theta TMS; Device: Arrhythmic TMS
- TMS to PMd followed by TMS to Mid-dlPFC (Experimental): Participants would receive TMS while performing a cognitive control task. In their first stimulation session, the TMS coil will be placed over PMd region on the scalp. In their second session, the TMS coil will be placed over the mid-dlPFC region on the scalp. During every session, participants receive Delta TMS (2.2 Hz), Theta TMS (6.5 Hz), and Arrhythmic TMS.
  Interventions: Device: Delta TMS; Device: Theta TMS; Device: Arrhythmic TMS

INTERVENTIONS:
Device: Delta TMS — TMS will be administered at the frequency of delta oscillation (2.2Hz)
  Other Names: MagPro X100 or R30 system
Device: Theta TMS — TMS will be administered at the frequency of theta oscillation (6.5Hz)
  Other Names: MagPro X100 or R30 system
Device: Arrhythmic TMS — TMS will be administered arrhythmically. In this intervention, the inter-pulse intervals are randomized between delta and theta durations for each trial, ensuring the same total number of pulses but without rhythmic consistency

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of rhythmic transcranial magnetic stimulation (TMS) delivered at delta (2.2 Hz) or theta (6.5 Hz) frequency on cognitive control.

This study aims to explore how targeted stimulation at delta and theta frequencies modulates brain activity to enhance cognitive performance in healthy populations.

DETAILED DESCRIPTION:
Neural oscillations are proposed to be a mechanism of coordinating information processing across distributed regions of cortex. Different neural oscillations may correspond to different underlying neural computations. Noninvasive brain stimulation allows experimenters to modulate specific neural oscillations by targeting particular frequency bands. Rhythmic transcranial magnetic stimulation (TMS) has been previously demonstrated to entrain neural oscillations at the frequency of stimulation.

Previous evidence suggests that cognitive control task paradigms elicit distinct activity in both Delta band (2-3 Hz) and Theta band (4-7 Hz). This task is designed to examine hierarchical cognitive control and includes two subtasks. In the Response Task, participants see a colored fixation cross and must make a button press with a specific finger. The stimulus to response mapping is memorized ahead of time. The number of stimulus to response rules is manipulated as four (low set-size) or eight (high set-size). In the Dimension Task, participants see two objects and must judge whether they are the same or different depending on one of two features. One feature is the shape of the object as either tall or wide. The other feature is the complexity of the objects as either being simple and smooth or complex and multifaceted. In this task, delta oscillations (2-3 Hz) are associated with rule abstraction, engaging the mid-dorsolateral prefrontal cortex (mid-dlPFC), while theta oscillations (4-7 Hz) are linked to stimulus-action associations and working memory load, with increased theta activity observed in the dorsal premotor area (PMd) under high set-size conditions.

For the current study, the investigators propose to deliver rhythmic trains of TMS in either delta frequency, theta frequency, or an arrhythmic control to modulate neural processing during a cognitive control task. By collecting simultaneous EEG with TMS, the investigators will be able to measure the entrained oscillations from rhythmic TMS. By applying delta frequency, theta frequency, and arrhythmic TMS during the performance of the task at each location, the investigators will be able to examine the causal relationship of delta oscillations at mid-dlPFC in rule abstraction and theta oscillations at PMd in stimulus-action associations. The stimulation is designed to enhance task performance by amplifying the neural activity patterns observed under these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 18 and 35.
* Must be able to provide informed consent.
* Must have normal or corrected-to-normal vision.
* Participants must be right-handed.
* Willingness to comply with all study procedures and availability for the study duration.
* Proficiency in speaking and understanding English.

Exclusion Criteria:

* Must not be color-blind
* Current treatment for ADHD/ADD.
* History of neurological disorders, including but not limited to the following specified conditions
* Epilepsy or seizures (excluding childhood febrile seizures).
* Dementia, Parkinson's disease, multiple sclerosis, cerebral aneurysm, or brain tumors.
* History of stroke or traumatic brain injury.
* Medical conditions or treatments that could interfere with study participation (e.g., unstable cardiac disease, HIV/AIDS, malignancy, or renal impairment).
* Prior brain surgery or presence of brain devices/implants (e.g., cochlear implants or aneurysm clips).
* Females who are pregnant or breastfeeding.
* Use of specific medications, including but not limited to ADHD medications or benzodiazepines, which may interfere with EEG measurements or task performance
* Any condition that, in the opinion of the investigator, increases risk or hinders full compliance with the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Change in Accuracy | Baseline (week 1); Session 1 (week 2); Session 2 (week 3)
  The Accuracy, reflecting the participants' ability to correctly follow task rules and make accurate judgments based on the given stimulus, is calculated as the percentage of correct responses across trials. The value range is 0% (no correct responses) to 100% (all responses correct), with a larger number denoting more correct responses.

SECONDARY OUTCOMES:
Change in Response Time | Baseline (week 1); Session 1 (week 2); Session 2 (week 3)
  The Response Time (RT), reflects the time taken by participants to respond to stimuli during the task. The value range is 0 seconds to 2 seconds, with a smaller number denoting faster responses.
Change in Amplitude of Neural Oscillations in mid-dlPFC | Baseline (week 1); Session 1 (week 2); Session 2 (week 3)
  The electrical activity of the brain is recorded during the performance of the task and brain stimulation. The investigators will perform Morlet wavelet convolution on the recorded electrical signal to calculate the amplitude of neural oscillations in the frequency bands: Delta (2-3 Hz) and Theta (4-7 Hz). The amplitude of neural oscillations is reported in the region that is being stimulated. The change in amplitude is normalized for each participant as the percent change from the amplitude during the baseline compared to the stimulation session (Session 1 or Session 2).
Change in Amplitude of Neural Oscillations in PMd | Baseline (week 1); Session 1 (week 2); Session 2 (week 3)
  The electrical activity of the brain is recorded during the performance of the task and brain stimulation. The investigators will perform Morlet wavelet convolution on the recorded electrical signal to calculate the amplitude of neural oscillations in the frequency bands: Delta (2-3 Hz) and Theta (4-7 Hz). The amplitude of neural oscillations is reported in the region that is being stimulated. The change in amplitude is normalized for each participant as the percent change from the amplitude during the baseline compared to the stimulation session (Session 1 or Session 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University Psychology Dept Bldg A411, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615